CLINICAL TRIAL: NCT00356434
Title: Study of Patient Compliance and Comfort Using Sequential Compression Devices and Foot Pumps for DVT Prevention
Brief Title: A Comparison of Sequential Compression Devices and Foot Pumps in the Obstetric Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI assigned to a different hospital;difficulty recruiting patients
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: foot pump vs SCD
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Thrombophilia
Keywords: deep vein thrombosis; thrombophilia; pregnancy; thromboprophylaxis; decreased mobility; hospitalization
MeSH Terms: conditions — Thrombophilia; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will have the Kendall, A-V foot impulse pump, model 6060 applied to their lower extremities to prevent DVT
  Interventions: Device: Kendall A-V foot impulse pump, model 6060
- 2 (Active Comparator): Patients will have the Kendall,sequential compression device, model 9525 applied to the lower extremities to prevent DVT
  Interventions: Device: Kendall sequential compression device, model 9525

INTERVENTIONS:
Device: Kendall A-V foot impulse pump, model 6060 — Will wear device for DVT prevention and receive questionnaire about compliance and comfort. Will also undergo random checks to confirm compliance with instructions and use
  Arms: 1
Device: Kendall sequential compression device, model 9525 — Will wear device for DVT prevention and receive questionnaire about compliance and comfort. Will also undergo random checks to confirm compliance with instructions and use
  Arms: 2

SUMMARY:
The researchers at Johns Hopkins University believe that the foot pump will be superior to sequential compression devices in comfort and patient compliance which may increase provider efforts to prevent deep vein thrombosis (DVT) in pregnancy.

DETAILED DESCRIPTION:
The investigators will be comparing sequential compression devices (SCDs) to foot pumps to determine if foot pumps will be better tolerated by obstetric patients, both antepartum and intrapartum. Patients in whom thromboembolic prophylaxis is deemed necessary and ordered by the treating physician, who agree to participate in the study will be randomly assigned to receive SCDs or the foot pump as part of their thromboembolic prophylaxis regimen. The investigators will administer a questionnaire to assess patients' satisfaction and comfort with each device and they will be asked to complete a log of hours they wore their assigned device for a 7 day period (or as long as they are prescribed). Random spot checks to verify compliance will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Bedrest
* Thrombophilia
* Prescribed DVT prophylaxis

Exclusion Criteria:

* Active DVT

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abimbola Aina, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986

RESULTS

PARTICIPANT FLOW:
Groups:
- Foot Pump: Patients will have the Kendall, A-V foot impulse pump, model 6060 applied to their lower extremities to prevent Deep Vein Thrombosis (DVT)
  Kendall A-V foot impulse pump, model 6060: Will wear device for DVT prevention and receive questionnaire about compliance and comfort. Will also undergo random checks to confirm compliance with instructions and use
- Sequential Compression Device: Patients will have the Kendall,sequential compression device, model 9525 applied to the lower extremities to prevent DVT
  Kendall sequential compression device, model 9525: Will wear device for DVT prevention and receive questionnaire about compliance and comfort. Will also undergo random checks to confirm compliance with instructions and use
Period: Overall Study
Arm/Group | Foot Pump | Sequential Compression Device
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Foot Pump: Patients will have the Kendall, A-V foot impulse pump, model 6060 applied to their lower extremities to prevent DVT
  Kendall A-V foot impulse pump, model 6060: Will wear device for DVT prevention and receive questionnaire about compliance and comfort. Will also undergo random checks to confirm compliance with instructions and use
- Total: Total of all reporting groups
Arm/Group | Foot Pump | Sequential Compression Device | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Comfort Level
Description: Scale of 1-10 (1 being very uncomfortable and 10 being very uncomfortable) describing level of comfort during the time of device use (composite score of heat, softness, discomfort).
Time Frame: once during first 7 days of hospitalization
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Foot Pump | Sequential Compression Device
Number analyzed (Participants) | 4 | 7
units on a scale | 7 [5 to 8] | 8 [6 to 10]

2. Primary Outcome: Patient Compliance
Description: Nurse conducting random checks throughout hospital stay and events of noncompliance will be recorded
Time Frame: for 1-7 days during hospitalization
Population: Data was not collected for this outcome measure, as the study was terminated prematurely.
Arm/Group | Foot Pump | Sequential Compression Device
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: DVT Prevention
Description: positive DVT on ultrasound
Time Frame: up to 3 months
Population: Data was not collected for this outcome measure, as the study was terminated prematurely.
Arm/Group | Foot Pump | Sequential Compression Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Foot Pump | Sequential Compression Device
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No